CLINICAL TRIAL: NCT06092138
Title: Edge Computing Platform for Spine Health Risk Management Based on IoT Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-NECKBRACE
Record Dates: First submitted 2023-09-27; First posted 2023-10-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cervical Disc Herniation; Cervical Spinal Stenosis; Ossification of Posterior Longitudinal Ligament; Neckbrace Device
Keywords: Rehabilitation; Neckbrace Device; Cervical Diesase
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wearable Device Group (Experimental): The Wearable Device Group uses wearable devices to perform rehabilitation exercises using the provided strategies. It includes the application of IoT technology to build a cloud platform combining software and hardware, using the spine sensors described in this project to collect behavioral data (it is recommended that they be worn during working hours every day for no less than 7 hours/week), and using end-to-end AI algorithms for health monitoring; the visualized data is synchronized to the spine health platform for real-time viewing and analysis by both doctors and patients. Through cell phone software and internet platform, spine health files are established to realize convenient and efficient communication between patients and professional doctors.
  Interventions: Device: Wearable Device
- Traditional group (No Intervention): The Traditional intervention group used traditional interventions, i.e., routine patient education, guidance on rehabilitation exercises, and tips on proper lifestyle habits.

INTERVENTIONS:
Device: Wearable Device — Whether to use wearable devices.
  Arms: Wearable Device Group

SUMMARY:
This project proposes to monitor the spinal posture of a person at rest and in motion in real time through a sensor device that contains spinal health monitoring as its core. By calibrating the five core planes on the spine and using AI algorithms to train the model, the relationship between the core plane data and spine health is established.This project will output medical-grade and consumer-grade wearable spine healthcare and monitoring products, establish an interactive platform to connect the wearer, the data terminal and the professional medical team, so that patients can easily get professional health advice and reminders during home healthcare and rehabilitation; and through the collection of spine health data, establish a national spine health database.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 60 years.
* Degenerative diseases of the cervical spine such as cervical disc herniation, cervical stenosis, ossification of the posterior longitudinal ligament, etc., but surgery is not considered for the time being.
* Available for clinical follow-up and agree to long-term clinical follow-up and sign informed consent.

Exclusion Criteria:

* Age less than 18 years or more than 60 years.
* Life expectancy less than 1 year.
* Suffering from severe dementia (MMSE score less than 18).
* Suffering from other serious medical conditions.
* Inability to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | Enrollment baseline，the first month, the second month, the third month
  Evaluate the efficacy of the device in reducing patients' pain. A score of 0 indicates no pain and a score of 10 represents the most severe pain that is unbearable.
neck disability index | Enrollment baseline，the first month, the second month, the third month
  The NDI consists of 10 items, including two parts: neck pain and related symptoms and activities of daily living. Each item has a minimum score of 0 and a maximum score of 5, with higher scores indicating more severe dysfunction.
quality of life short form 12 | Enrollment baseline，the first month, the second month, the third month
  Evaluate the efficacy of the device in improving patients' quality of life.The maximum value of physical score is 56.58 and the maximum value of mental score is 60.76. A higher score indicates a better quality of life.

SECONDARY OUTCOMES:
Change in muscle strength (grade) | Enrollment baseline, the third month
  Change in muscle strength (grade) = Muscle strength at the third month - Muscle strength at enrollment.
  Muscle strength is graded from 0 to 5, with higher grades indicating better motor function of the extremities.
  Muscle strength is evaluated by experienced physicians.
Change in muscle tone (grade) | Enrollment baseline, the third month
  Change in muscle tone (grade) = Muscle tone at enrollment -Muscle tone at the third month.
  Muscle tone is graded into 6 grades, with higher grades indicating worse motor function of the extremities.
  Muscle tone is evaluated by experienced physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Edge Computing Platform for Spine Health Risk Management, Beijing, Beijing Municipality, China